CLINICAL TRIAL: NCT02410837
Title: NAVIGATE: Clinical Evaluation of superDimension™ Navigation System for Electromagnetic Navigation Bronchoscopy™
Status: Completed | Type: Observational
Sponsor: Medtronic - MITG (Industry)
Responsible Party: Sponsor
Other Study IDs: COVENBP0475
Record Dates: First submitted 2015-03-31; First posted 2015-04-08 (Estimated); Results first posted 2021-03-11 (Actual); Last update posted 2021-05-10 (Actual); Status verified 2021-05

CONDITIONS: Lung Lesion(s) Requiring Evaluation
Keywords: lung lesion; biopsy; bronchoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years

INTERVENTIONS:
Procedure: Electromagnetic Navigation Bronchoscopy
  Other Names: ENB; superDimension

SUMMARY:
The purpose of this study is to evaluate outcomes following electromagnetic navigation bronchoscopy™ (ENB™) procedures using the superDimension™ navigation system.

DETAILED DESCRIPTION:
This clinical trial information was submitted voluntarily under the applicable law and, therefore, certain submission deadlines may not apply. (That is, clinical trial information for this applicable clinical trial was submitted under section 402(j)(4)(A) of the Public Health Service Act and 42 CFR 11.60 and is not subject to the deadlines established by sections 402(j)(2) and (3) of the Public Health Service Act or 42 CFR 11.24 and 11.44.)

ELIGIBILITY:
Inclusion Criteria:

* Subject presents with lung lesion(s) requiring evaluation
* Subject is willing and able to provide informed consent to participate in the study
* Subject is candidate for elective ENB™ procedure
* Subject is over the age of 18

Exclusion Criteria:

* The subject is unable or unwilling to comply with study follow-up schedule
* The subject has participated in an investigational drug or device research study within 30 days of enrollment that would interfere with this study
* Female subjects who are pregnant or nursing as determined by standard site practices

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects that meet the various inclusion/exclusion criteria will be enrolled consecutively by each participating site.
Sampling Method: Non-Probability Sample
Enrollment: 1388 (Actual)
Dates: Start 2015-04-16 (Actual); Primary Completion 2019-11-01 (Actual); Study Completion 2019-11-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sandeep Khandhar, MD, Principal Investigator — Inova Fairfax Hospital; Erik Folch, MD, Principal Investigator — Massachusetts General Hospital
Locations (37):
- United States (29):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Pulmonary Associates of Mobile, P.C., Mobile, Alabama
  - Palo Alto Medical Foundation, Mountain View, California
  - Pulmonary and Sleep of Tampa Bay, Brandon, Florida
  - Ocala Lung and Critical Care, Ocala, Florida
  - Cancer Treatment Centers of America, Newnan, Georgia
  - The University of Chicago, Chicago, Illinois
  - Pulmonary and Critical Care Associates of Baltimore, Baltimore, Maryland
  - University of Michigan Health Systems, Ann Arbor, Michigan
  - Virtua Medical Group, PA, Marlton, New Jersey
  - University of Rochester, Rochester, New York
  - Carolina's Healthcare System, Charlotte, North Carolina
  - Duke University, Durham, North Carolina
  - East Carolina University, Greenville, North Carolina
  - Pinehurst Medical Center, Pinehurst, North Carolina
  - University of Cincinnati Physicians Company LLC, Cincinnati, Ohio
  - University Hospitals of Case Medical Center, Cleveland, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Penn Highlands Healthcare, DuBois, Pennsylvania
  - UPMC - Shadyside Medical Center, Pittsburgh, Pennsylvania
  - Pulmonary Medicine Center of Chattanooga - Memorial Health, Chattanooga, Tennessee
  - Blount Memorial Hospital, Maryville, Tennessee
  - Vanderbilt University, Nashville, Tennessee
  - Seton Medical Center Austin, Austin, Texas
  - East Texas Medical Center, Tyler, Texas
  - Providence Health Center, Waco, Texas
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Charleston Area Medical Center, Charleston, West Virginia
  - Gundersen Lutheran Medical Foundation, Inc, La Crosse, Wisconsin
- Austria (2):
  - AKH Linz, Linz
  - Salzburger Landesklinik (SALK), Salzburg
- Rigshospitalet - Copenhagen, Copenhagen, Denmark
- University Hospitals of Saint Etienne France, Saint-Etienne, France
- Italy (2):
  - Azienda Ospedaliero Universitaria Careggi, Florence
  - IRCCS Azienda Ospedaliera Universitaria San Martino - IST, Genova
- Hospital Fundacion Jimenez Diaz, Madrid, Spain
- St. Bartholomew's Hospital, London, United Kingdom

REFERENCES:
- [Derived] Bowling MR, Folch EE, Khandhar SJ, Kazakov J, Krimsky WS, LeMense GP, Linden PA, Murillo BA, Nead MA, Pritchett MA, Teba CV, Towe CW, Williams T, Anciano CJ. Fiducial marker placement with electromagnetic navigation bronchoscopy: a subgroup analysis of the prospective, multicenter NAVIGATE study. Ther Adv Respir Dis. 2019 Jan-Dec;13:1753466619841234. doi: 10.1177/1753466619841234. PMID 30958102
- [Derived] Khandhar SJ, Bowling MR, Flandes J, Gildea TR, Hood KL, Krimsky WS, Minnich DJ, Murgu SD, Pritchett M, Toloza EM, Wahidi MM, Wolvers JJ, Folch EE; NAVIGATE Study Investigators. Electromagnetic navigation bronchoscopy to access lung lesions in 1,000 subjects: first results of the prospective, multicenter NAVIGATE study. BMC Pulm Med. 2017 Apr 11;17(1):59. doi: 10.1186/s12890-017-0403-9. PMID 28399830
- [Derived] Folch EE, Bowling MR, Gildea TR, Hood KL, Murgu SD, Toloza EM, Wahidi MM, Williams T, Khandhar SJ. Design of a prospective, multicenter, global, cohort study of electromagnetic navigation bronchoscopy. BMC Pulm Med. 2016 Apr 26;16(1):60. doi: 10.1186/s12890-016-0228-y. PMID 27113209

RESULTS

PARTICIPANT FLOW:
Groups:
- NAVIGATE (Single Arm Study): Observational NAVIGATE arm (single arm study, no comparator)
Period: Overall Study
Arm/Group | NAVIGATE (Single Arm Study)
Started | 1388
Procedure | 1388
1-Month | 1374
12-Month | 1121
24-Month | 900
Completed | 900
Not Completed | 488
Not completed — Death | 387
Not completed — Lost to Follow-up | 50
Not completed — Withdrawal by Subject | 44
Not completed — Physician Decision | 6
Not completed — Moved to nursing home, cannot communicat | 1

BASELINE CHARACTERISTICS:
Population: 1388 subjects were enrolled. 1329 subjects had an indication for procedure for lesion biopsy. 1260 subjects had procedure for biopsy with successful navigation. 1529 is the number of lesions for biopsy.
Units Other Than Participants: Number of Lesions for Biopsy
Arm/Group | NAVIGATE (Single Arm Study)
Number analyzed (Participants) | 1388
Number analyzed (Number of Lesions for Biopsy) | 1529
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 494
  >=65 years | 894
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.6 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 698
  Male | 690
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 95
  Not Hispanic or Latino | 1268
  Unknown or Not Reported | 25
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: American Indian or Alaska Native | 4
  Race: Asian | 8
  Race: Native Hawaiian or Other Pacific Islander | 1
  Race: Black or African American | 164
  Race: White | 1162
  Race: Other | 2
  Race: Unknown | 10
  Race: Unable to report | 37
Region of Enrollment [Number; unit: participants]
  Austria | 20
  United States | 1213
  Denmark | 24
  Italy | 36
  United Kingdom | 42
  France | 3
  Spain | 50
Tobacco history (current or former) [Count of Participants; unit: Participants] | 1107
Chronic obstructive pulmonary disease [Count of Participants; unit: Participants] | 601
Personal history of cancer [Count of Participants; unit: Participants] | 667
Family history of cancer [Count of Participants; unit: Participants] | 816
General anesthesia [Count of Participants; unit: Participants] | 1086
Radial Endobronchial Ultrasound (R-EBUS) used during Electromagnetic Navigation Bronchoscopy (ENB) [Count of Participants; unit: Participants] | 703
Cone-beam Computed Tomography (CBCT) used during ENB [Count of Participants; unit: Participants] | 77
Fluoroscopy used during ENB [Number; unit: number of lesions] — Population: Number of lesions (subjects could have more than one lesion)
  number of lesions | 1299
Rapid on-site evaluation (ROSE) used [Count of Participants; unit: Participants] — Population: Number of subjects undergoing ENB for lesion biopsy where navigation was successful
  Participants
    number analyzed (Participants) | 1260
    (all) | 777
Average number of lesions biopsied per subject [Mean (Standard Deviation); unit: Number of lesions] — Population: 1329 subjects who underwent ENB for lung lesion biopsy
  Number of lesions
    number analyzed (Participants) | 1329
    (all) | 1.2 (0.4)
Lesion size (mm) [Median (Inter-Quartile Range); unit: millimeters] — There were 1529 lesions in the study. 1528 reported measurement on lesion size. Population: Number of lesions where size was provided
  millimeters | 20.0 [14.0 to 29.0]
Upper lobe lesion location [Number; unit: number of lesions] — Population: Number of lesions (subjects could have more than one lesion)
  number of lesions | 897
Peripheral third of the lung [Number; unit: number of lesions] — Population: Number of lesions (subjects could have more than one lesion)
  number of lesions | 1036
Lesion distance to pleura (mm) [Median (Inter-Quartile Range); unit: millimeters] — Population: Number of lesions where distance was provided. 1514 lesions in 1317 subjects had "lesion distance to pleura" information.
  millimeters
    number analyzed (Participants) | 1317
    number analyzed (Number of Lesions for Biopsy) | 1514
    (all) | 9.0 [0.0 to 20.0]
Pure to mostly ground glass opacity (GGO) lesions (Suzuki Class 1 or 2) [Number; unit: participants] — Population: Number of lesions where ground glass was evaluated. 1523 lesions in 1323 subjects where ground glass opacity (GGO) was evaluated.
  participants
    number analyzed (Participants) | 1323
    number analyzed (Number of Lesions for Biopsy) | 1523
    (all) | 95
Spiculated lesion border [Number; unit: participants] — Population: Number of lesions where lesion border was evaluated and reported. 1527 lesions in 1328 subjects had lesion border information.
  participants
    number analyzed (Participants) | 1328
    number analyzed (Number of Lesions for Biopsy) | 1527
    (all) | 923
Bronchus sign present on Computed Tomography (CT) [Number; unit: participants] — Population: Number of lesions where bronchus sign presence was evaluated
  participants | 777
Pre-test probability of malignancy >65% (Physician Estimate) [Number; unit: number of lesions] — Population: Number of lesions where the physicians estimate of pre-test probability of malignancy was evaluated
  number of lesions
    number analyzed (Participants) | 1027
    number analyzed (Number of Lesions for Biopsy) | 1188
    (all) | 730

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Pneumothorax (Grade 2+)
Description: The primary endpoint is the incidence of pneumothorax related to the ENB™ index procedure rated as Grade 2 or higher according to the Common Terminology Criteria for Adverse Events (CTCAE) scale.
  Pneumothorax is a disorder characterized by abnormal presence of air in the pleural cavity resulting in the collapse of the lung.
  Severity increases as grade increases. Grade 1: Asymptomatic; clinical or diagnostic observations only; intervention not indicated; Grade 2: Symptomatic; intervention indicated (e.g., tube placement without sclerosis); Grade 3: Sclerosis and/or operative intervention indicated; hospitalization indicated; Grade 4: Life-threatening consequences; urgent intervention indicated; Grade 5: Death
Time Frame: index procedure visit
Population: All subjects included in this analysis
Measure: Count of Participants; unit: Participants
Arm/Group | NAVIGATE (Single Arm Study)
Number analyzed (Participants) | 1388
Participants | 44

2. Secondary Outcome: Incidence of Pneumothorax (All)
Description: The incidence of pneumothorax related to all ENB™ index procedures will be evaluated.
Time Frame: index procedure visit
Measure: Count of Participants; unit: Participants
Arm/Group | NAVIGATE (Single Arm Study)
Number analyzed (Participants) | 1388
Participants | 65

3. Secondary Outcome: Incidence of Bronchopulmonary Hemorrhage
Description: The incidence of bronchopulmonary hemorrhage (rated as Grade 2 or higher according to th CTCAE scale) related to all ENB™ index procedures will be evaluated.
  Bronchopulmonary hemorrhage is a disorder characterized by bleeding from the bronchial wall and/or lung parenchyma.
  Severity increases as grade increases. Grade 1: Mild symptoms; intervention not indicated; Grade 2: Moderate symptoms; medical intervention indicated; Grade 3: Transfusion, radiologic, endoscopic, or operative intervention indicated (e.g., hemostasis of bleeding site); Grade 4: Life-threatening respiratory or hemodynamic compromise; intubation or urgent intervention indicated; Grade 5: Death
Time Frame: index procedure visit
Measure: Count of Participants; unit: Participants
Arm/Group | NAVIGATE (Single Arm Study)
Number analyzed (Participants) | 1388
Participants | 23

4. Secondary Outcome: Incidence of Respiratory Failure
Description: The incidence of respiratory failure (rated as Grade 4 or higher according to the CTCAE scale) related to all ENB™ index procedures will be evaluated.
  A respiratory failure is a disorder characterized by impaired gas exchange by the respiratory system resulting in hypoxemia and a decrease in oxygenation of the tissues that may be associated with an increase in arterial levels of carbon dioxide.
  Severity increases as grade increases. Within CTCAE, there are no grades 1, 2, or 3 for Respiratory Failure.
  Grade 4: Life-threatening consequences; urgent intervention, intubation, or ventilatory support indicated; Grade 5: Death
Time Frame: index procedure visit
Measure: Count of Participants; unit: Participants
Arm/Group | NAVIGATE (Single Arm Study)
Number analyzed (Participants) | 1388
Participants | 8

5. Secondary Outcome: Quality of Life (Mobility, Self-care, Activities, Pain/Discomfort, Anxiety/Depression, Health State)
Description: Subject health status evaluated by EuroQol-5d (EQ-5D) questionnaire at all visits. (Mobility, Self-care, Activities, Pain/Discomfort, Anxiety/Depression, Health state) Questionnaire from EuroQol Group. Outcome reported on overall health state over time. 0 = worst imaginable health state, 100 = best imaginable health state.
Time Frame: Baseline, 1 month, 12 month, and 24 month follow up visits
Population: Number of subjects who completed the EQ-5D at the baseline visit.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | NAVIGATE (Single Arm Study)
Number analyzed (Participants) | 1364
score on a scale
  Baseline | 70.2 (19.4)
  1-Month: number analyzed (Participants) | 1225
  1-Month | 69.2 (20.4)
  12-Month: number analyzed (Participants) | 927
  12-Month | 70.0 (20.6)
  24-Month: number analyzed (Participants) | 798
  24-Month | 72.6 (18.7)

6. Secondary Outcome: Subject Satisfaction
Description: Subject satisfaction evaluation at the 1 month visit.
  The question was "overall, how satisfied were you with the ENB procedure". Options were:
  1. Totally Dissatisfied
  2. Dissatisfied
  3. Neutral
  4. Satisfied
  5. Extremely Satisfied
Time Frame: at the 1 month follow up visit
Population: Subjects who completed the 1-month subject satisfaction questionnaire (How satisfied are you with ENB on a scale of 1-5)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | NAVIGATE (Single Arm Study)
Number analyzed (Participants) | 1227
score on a scale | 4.4 (0.8)

7. Secondary Outcome: Subject Productivity and Activity
Description: Electromagnetic Navigation Bronchoscopy (ENB) procedure effect on subject productivity and activity using the ENB Productivity and Activity Questionnaire (ENB-PAQ) will be evaluated.
  The outcome measurement is the effect of ENB on their regular daily activities on a scale of 0-10 (0=no effect, 10=completely prevented).
Time Frame: at the 1 month follow up visit
Population: Number of subjects who completed the ENB-PAQ at 1-month
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | NAVIGATE (Single Arm Study)
Number analyzed (Participants) | 854
score on a scale | 0.9 (2.1)

8. Secondary Outcome: Diagnostic Yield
Description: Diagnostic yield will be evaluated for all ENB™ index procedures performed for suspicion of cancer or other lung diseases in a lung lesion.
  Diagnostic yield was calculated per subject as the rate of true positives (TP) (for malignancy) plus true negatives (TN) (for malignancy) out of all subjects with attempted lung lesion biopsies (the denominator included subjects with no tissue obtained due to unsuccessful navigation).
Time Frame: up to 24 months
Population: Per subject including all those with attempted lung lesion biopsies. This includes any with unsuccessful navigation, but excludes subjects with insufficient follow-up where True Positive, True Negative, False Positive and False Negative could not be determined by 24 months.
Measure: Count of Participants; unit: Participants
Arm/Group | NAVIGATE (Single Arm Study)
Number analyzed (Participants) | 1212
Participants | 822

9. Secondary Outcome: Sensitivity
Description: Sensitivity will be evaluated for all ENB™ index procedures performed for suspicion of cancer or other lung diseases in a lung lesion. [True Positives =TP, False Negatives = FN].
  (TP / [TP+FN])
Time Frame: up to 24 months
Population: Number of subjects with a True Positive (TP) for Malignancy or False Negative (FN) for Malignancy diagnosis by 24-months.
Measure: Count of Participants; unit: Participants
Arm/Group | NAVIGATE (Single Arm Study)
Number analyzed (Participants) | 858
Participants | 537

10. Secondary Outcome: Specificity
Description: Specificity will be evaluated for all ENB™ index procedures performed for suspicion of cancer or other diseases in a lung lesion. [True Negatives = TN, False Positives = FN] (TN / [FP+TN])
Time Frame: up to 24 months
Population: Number of subjects with a False Positive (FP) for Malignancy or True Negative (TN) for Malignancy diagnosis by 24-months.
Measure: Count of Participants; unit: Participants
Arm/Group | NAVIGATE (Single Arm Study)
Number analyzed (Participants) | 285
Participants | 285

11. Secondary Outcome: Positive Predictive Value
Description: Positive predictive value (PPV) will be evaluated for all ENB™ index procedures performed for suspicion of cancer or other diseases in a lung lesion. [True Positives = TP, False Positives = FP] (TP / [TP+FP])
Time Frame: up to 24 months
Population: Number of subjects with a True Positive (TP) for Malignancy or False Positive (FP) for Malignancy diagnosis by 24-months.
Measure: Count of Participants; unit: Participants
Arm/Group | NAVIGATE (Single Arm Study)
Number analyzed (Participants) | 537
Participants | 537

12. Secondary Outcome: Negative Predictive Value
Description: Negative Predictive Value (NPV) will be evaluated for all ENB™ index procedures performed for suspicion of cancer or other diseases in a lung lesion. [True Negatives = TN, False Negatives = FN] (TN / [FN+TN])
Time Frame: up to 24 months
Population: Number of subjects with a False Negative (FN) for Malignancy or True Negative (TN) for Malignancy diagnosis by 24-months.
Measure: Count of Participants; unit: Participants
Arm/Group | NAVIGATE (Single Arm Study)
Number analyzed (Participants) | 606
Participants | 285

13. Secondary Outcome: Repeat Biopsy Rate
Description: Repeat biopsy rate due to lack of diagnosis during the ENB™ index procedure will be evaluated for all ENB™ index procedures performed for suspicion of cancer or other diseases in a lung lesion.
Time Frame: up to 24 months
Population: Number of subjects with navigation complete and tissue obtained
Measure: Count of Participants; unit: Participants
Arm/Group | NAVIGATE (Single Arm Study)
Number analyzed (Participants) | 1260
Participants | 334

14. Secondary Outcome: Tissue Adequacy for Molecular Genetic Testing
Description: Tissue adequacy for molecular genetic testing (if applicable).
Time Frame: at index procedure visit
Population: This is the number of lesions diagnosed with primary lung adenocarcinoma or non-small-cell lung cancer not otherwise specified, where molecular genetic testing was attempted. This does not include all lesions biopsied as not all lesions had one of these specific diagnoses, nor did all these with these specific diagnoses have molecular testing attempted.
Measure: Count of Units; unit: Lesions
Units Other Than Participants: Lesions
Arm/Group | NAVIGATE (Single Arm Study)
Number analyzed (Participants) | 102
Number analyzed (Lesions) | 110
Lesions | 89

15. Secondary Outcome: Diagnosis
Description: Diagnosis will be evaluated for all ENB™ index procedures performed for suspicion of cancer or other diseases in a lung lesion (per subject)
Time Frame: up to 24 months
Population: Number of subjects where navigation was complete and tissue was obtained for a diagnosis. Subjects with multiple lesion diagnoses may be represented more than once in all subcategories.
Measure: Count of Units; unit: Diagnoses
Units Other Than Participants: Diagnoses
Arm/Group | NAVIGATE (Single Arm Study)
Number analyzed (Participants) | 1260
Number analyzed (Diagnoses) | 1276
Diagnoses
  Adenocarcinoma | 279
  Squamous Carcinoma | 133
  Other Non-small cell lung cancer | 16
  Small cell carcinoma | 26
  Neuroendocrine Carcinoma | 17
  Metastatic Carcinoma | 49
  Lymphoma | 2
  Malignant Cells (unable to characterize) | 12
  Malignant Atypical Cells | 3
  Other Malignancy | 3
  Benign Inflammation | 198
  Benign Other | 97
  Inconclusive | 201
  Normal Lung Tissue | 119
  Hamartoma | 1
  Granuloma | 20
  Bacterial Infection | 24
  Fungal Infection | 14
  Viral Infection | 3
  Organizing Pneumonia | 7
  Interstitial Lung Disease | 7
  Lymphocytes | 10
  Benign Atypical Cells | 20
  Other Benign | 15

16. Secondary Outcome: Stage at Diagnosis
Description: Stage at diagnosis (if applicable) will be evaluated for all ENB™ index procedures performed for suspicion of cancer or other diseases in a lung lesion. (Diagnosis worsens as stage number increases).
  Refer to the American Joint Committee on Cancer, 7th edition on Lung Cancer Staging. A brief description is provided here.
  Stage I = small lesions, no lymph node involvement Stage II = larger lesions and/or lymph nodes on sides of lung involved Stage III = larger lesions and/or lymph nodes in middle of chest involved Stage IV = metastases to other organs
Time Frame: up to 24 months
Population: Number of subjects diagnosed with primary lung cancer.
Measure: Count of Participants; unit: Participants
Arm/Group | NAVIGATE (Single Arm Study)
Number analyzed (Participants) | 468
Participants
  Stage I | 251
  Stage II | 52
  Stage III | 81
  Stage IV | 84

17. Secondary Outcome: Success Rate of Accurate Placement of Fiducial Markers
Description: The success rate of accurate placement of fiducial markers demonstrated through follow up imaging will be evaluated for all ENB™ index procedures conducted for placement of fiducial markers.
Time Frame: at index procedure visit
Population: Number of subjects where ENB was used to aid in placement of fiducial markers, and follow-up imaging data was available.
Measure: Count of Participants; unit: Participants
Arm/Group | NAVIGATE (Single Arm Study)
Number analyzed (Participants) | 269
Participants | 253

18. Secondary Outcome: Success Rate of Dye Marking
Description: The success rate of dye marking demonstrated by successful surgical resection will be evaluated for all ENB™ index procedures conducted for dye marking in preparation for surgical resection.
Time Frame: at index procedure visit
Population: Number of subjects where ENB was used to aid in pleural dye marking.
Measure: Count of Participants; unit: Participants
Arm/Group | NAVIGATE (Single Arm Study)
Number analyzed (Participants) | 23
Participants | 21

19. Secondary Outcome: Success Rate of Obtaining Lymph Node Biopsy
Description: The success rate of obtaining a lymph node biopsy to provide the stage of diagnosis will be evaluated for all ENB™ index procedures conducted for a lymph node biopsy.
Time Frame: at index procedure visit
Population: Number of subjects where ENB was used to aid in lymph node biopsy.
Measure: Count of Participants; unit: Participants
Arm/Group | NAVIGATE (Single Arm Study)
Number analyzed (Participants) | 36
Participants | 31

ADVERSE EVENTS:
Time Frame: Up to 24 months post procedure
Description: ISO 14155 event definitions were used. The following AEs were required to be reported:
  All AEs related to the superDimension™ navigation system, associated tools, or ENB™ procedure (both index and any subsequent repeat ENB™ procedure); All deaths (all-cause); All pneumothoraces (all-cause); All bronchopulmonary hemorrhages (all-cause); All respiratory failures (all cause) Important note: not all events reported in the study were related to the study procedure or study device.
Arm/Group | NAVIGATE (Single Arm Study)
All-Cause Mortality (participants affected / at risk) | 403/1388
Serious Adverse Events (participants affected / at risk) | 497/1388
Other Adverse Events (participants affected / at risk) | 96/1388
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NAVIGATE (Single Arm Study) (N=1388)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 1 (1)
Cardiac arrest (Cardiac disorders) | 9 (9)
Cardiac failure (Cardiac disorders) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 3 (3)
Cardio-respiratory arrest (Cardiac disorders) | 16 (16)
Cardiopulmonary failure (Cardiac disorders) | 3 (3)
Cor pulmonale acute (Cardiac disorders) | 1 (1)
Left ventricular failure (Cardiac disorders) | 3 (3)
Myocardial infarction (Cardiac disorders) | 2 (2)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 (2)
Inguinal hernia (Gastrointestinal disorders) | 1 (1)
Intestinal infarction (Gastrointestinal disorders) | 1 (1)
Intestinal perforation (Gastrointestinal disorders) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1)
Death (General disorders) | 86 (86)
Disease progression (General disorders) | 2 (2)
Multiple organ dysfunction syndrome (General disorders) | 1 (1)
Acute hepatic failure (Hepatobiliary disorders) | 1 (1)
Cirrhosis alcoholic (Hepatobiliary disorders) | 1 (1)
Hepatorenal syndrome (Hepatobiliary disorders) | 1 (1)
Bacteraemia (Infections and infestations) | 1 (1)
Bacterial sepsis (Infections and infestations) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 7 (7)
Pneumonia fungal (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 5 (5)
Septic shock (Infections and infestations) | 2 (2)
Transmission of an infectious agent via product (Infections and infestations) | 1 (1)
Gun shot wound (Injury, poisoning and procedural complications) | 1 (1)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Procedural pneumothorax (Injury, poisoning and procedural complications) | 3 (3)
Failure to thrive (Metabolism and nutrition disorders) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1)
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Brain neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4)
Breast cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Extranodal marginal zone B-cell lymphoma (MALT type) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Leiomyosarcoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 18 (18)
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 23 (23)
Lung carcinoma cell type unspecified stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Lung carcinoma cell type unspecified stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 45 (45)
Lung squamous cell carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Lung squamous cell carcinoma stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Meningioma malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Metastatic pulmonary embolism (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Metastatic renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Metastatic uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3)
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3)
Non-small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Oesophageal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Oesophageal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4)
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Pharyngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Renal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3)
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (5)
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Uterine leiomyosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Cerebral infarction (Nervous system disorders) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 4 (4)
Goodpasture's syndrome (Renal and urinary disorders) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 8 (8)
Apnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Mediastinal haematoma (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 81 (83)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 15 (15)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 111 (138)
Arteriosclerosis (Vascular disorders) | 1 (1)
Arteriovenous fistula (Vascular disorders) | 1 (1)
Peripheral circulatory failure (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NAVIGATE (Single Arm Study) (N=1388)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 72 (73)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 24 (24)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institution and Investigator shall not publish the Study results until after Sponsor's multi-site publication of complete and final study results or until the elapse of twelve (12) months from the close of the Study at all Study sites, whichever occurs earlier; unless approved by Sponsor.

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2015-11-17): https://cdn.clinicaltrials.gov/large-docs/37/NCT02410837/Prot_SAP_ICF_000.pdf